CLINICAL TRIAL: NCT03400306
Title: A Phase 1, Single-Dose, Open-Label, Randomized Cross-Over Study Evaluating the Bioavailability and Food Effect of Veliparib Tablets Followed by an Extension in Subjects With Ovarian Cancer
Brief Title: A Study Evaluating the Bioavailability and Food Effect of Veliparib Tablets Followed by an Extension in Subjects With Ovarian Cancer
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Strategic considerations
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: M15-536; 2018-000313-20 (EudraCT Number)
Expanded Access: NCT03123211 (No longer available)
Record Dates: First submitted 2018-01-12; First posted 2018-01-17 (Actual); Last update posted 2021-12-08 (Actual); Status verified 2021-12

CONDITIONS: Cancer - Ovarian
Keywords: Cancer - Ovarian cancer; Bioavailability; Pharmacokinetics; Bioequivalence
MeSH Terms: conditions — Ovarian Neoplasms | interventions — veliparib; Capsules; Carboplatin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Part 1, Bioequivalence Sequence Group 1 (Experimental): Veliparib 400-mg doses administered orally on Day 1 of each 2-3 day period in Part 1 with the following sequence for the 3 dosing days: four 100 mg capsules under fasting conditions, followed by one 400-mg tablet under fasting conditions, then one 400 mg tablet under non-fasting conditions.
  Interventions: Drug: Veliparib, capsule; Drug: Veliparib, tablet
- Part 2, Extension (Experimental): Veliparib as monotherapy or in combination with carboplatin and paclitaxel, per investigators' discretion.
  Interventions: Drug: Veliparib, capsule; Drug: Carboplatin; Drug: Paclitaxel
- Part 1, Bioequivalence Sequence Group 2 (Experimental): Veliparib 400-mg doses administered orally on Day 1 of each 2-3 day period in Part 1 with the following sequence for the 3 dosing days: one 400-mg tablet under fasting conditions, followed by four 100 mg capsules under fasting conditions, then one 400 mg tablet under non-fasting conditions.
  Interventions: Drug: Veliparib, capsule; Drug: Veliparib, tablet

INTERVENTIONS:
Drug: Veliparib, capsule — capsule; 50 mg or 100 mg
  Other Names: ABT-888
Drug: Veliparib, tablet — tablet; 400 mg
  Other Names: ABT-888
  Arms: Part 1, Bioequivalence Sequence Group 1; Part 1, Bioequivalence Sequence Group 2
Drug: Carboplatin — Intravenous
  Other Names: Paraplatin
  Arms: Part 2, Extension
Drug: Paclitaxel — Intravenous
  Other Names: Taxol
  Arms: Part 2, Extension

SUMMARY:
This study will evaluate the bioavailability between the veliparib tablet formulation to the capsule formulation; and will assess the effect of food on veliparib bioavailability in participants with ovarian cancer.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of epithelial ovarian, fallopian tube, or primary peritoneal carcinoma.
* Laboratory values meeting protocol-specified criteria, including hematologic, kidney and liver function.
* Life expectancy of 12 weeks or greater.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2.
* Able to swallow and retain oral medication.
* Discontinued anti-cancer therapy and biological agent for antineoplastic intent 21 days prior to the first dose of study drug, not have undergone major surgery 28 days prior to the first dose of study drug; and have recovered to Grade 0 - 2 for any clinical significant adverse event effect(s)/toxicity(s) from previous therapy.
* Non-childbearing potential.

Exclusion Criteria:

* History or active medical condition(s) affecting absorption or motility or any surgical procedure that might interfere with gastrointestinal motility, pH or absorption.
* Evidence of refractory ascites.
* Has clinically relevant or significant electrocardiogram abnormalities.

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-11-15 (Estimated); Primary Completion 2021-11-16 (Actual); Study Completion 2021-11-16 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) | Up to approximately 8 days after initial dose of study drug
  Maximum observed plasma concentration (Cmax)
Time to Maximum Observed Plasma Concentration (Tmax) | Up to approximately 8 days after initial dose of study drug
  Time to maximum observed plasma concentration (Tmax).
Apparent Terminal Phase Elimination Rate Constant (β or Beta) | Up to approximately 8 days after initial dose of study drug
  Apparent terminal phase elimination rate constant (β or Beta).
Terminal Phase Elimination Half-life (t1/2) | Up to approximately 8 days after initial dose of study drug
  Terminal phase elimination half-life (t1/2)
Area Under the Plasma Concentration-time Curve (AUC) from Time 0 to Time of the Last Measurable Concentration (AUCt) | Up to approximately 8 days after initial dose of study drug
  Area under the plasma concentration-time curve (AUC) from time 0 to time of the last measurable concentration (AUCt).
AUC from time 0 to infinite time (AUC∞) | Up to approximately 8 days after initial dose of study drug
  AUC from time 0 to infinite time (AUC∞)

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie

IPD SHARING:
Plan to Share IPD: No